CLINICAL TRIAL: NCT03276806
Title: Capitalizing on Hospitalization to Engage Low SES Smokers in LDCT Screening: A Randomized Controlled Trial
Brief Title: Inpatient Smokers and LDCT Screening RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: American Lung Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-36854; LCD-507875 (Other Grant/Funding Number: American Lung Association)
Record Dates: First submitted 2017-09-05; First posted 2017-09-08 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Lung Cancer; Shared Decision Making
Keywords: CT low dose; nurse led intervention; safety net hospital; lung cancer screening with CTLD
MeSH Terms: conditions — Lung Neoplasms | interventions — SDM; Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDM + decision aid + tobacco counseling (Experimental): Participants will receive tobacco dependence/smoking cessation counseling by a nurse, SDM and a decision aid.
  Interventions: Behavioral: tobacco dependence/smoking cessation counseling; Behavioral: SDM; Other: Decision Aid
- LDCT brochure + tobacco counseling (Active Comparator): Participants will receive tobacco dependence/smoking cessation counseling by a nurse and a LDCT informational brochure.
  Interventions: Behavioral: tobacco dependence/smoking cessation counseling; Other: LDCT brochure

INTERVENTIONS:
Behavioral: tobacco dependence/smoking cessation counseling — Standard of care tobacco dependence/smoking cessation counseling offered to all smokers at Boston Medical Center.
Behavioral: SDM — SDM is three-fold to: 1) conduct a tailored discussion on tradeoffs of LDCT screening, consistent with CMS requirements for SDM using a decision aid; 2) directly connect interested patients to LDCT screening; 3) to empower and motivate patients to quit smoking within the LDCT screening context.
  Other Names: Shared decision making
  Arms: SDM + decision aid + tobacco counseling
Other: Decision Aid — The decision aid is a 4-page paper format with the following features: 1) LDCT screening harms and benefits information, written in plain language and using pictographs, easily understood by those with low health literacy; 2) prompts to clarify patient values and preferences and to stimulate discussion about trade-offs; 3) clear quit smoking messaging and resources (1-800-QUIT-NOW).
  Arms: SDM + decision aid + tobacco counseling
Other: LDCT brochure — A informational brochure developed by the BMC screening program about low dose CT screening for lung cancer.
  Arms: LDCT brochure + tobacco counseling

SUMMARY:
Current smokers who undergo annual low dose CT (LDCT) lung cancer screening and successfully quit smoking derive the greatest reduction in lung cancer mortality. Unfortunately, those at highest risk of lung cancer death- those with low socioeconomic status, blacks, and current smokers- are the same individuals that typically have reduced access to preventive healthcare such as smoking cessation services and screening tests. Furthermore, patients from underserved communities often have lower health literacy, less awareness of lung cancer screening, and a poor understanding of the trade-offs of LDCT screening. In 2015 the Center for Medicare and Medicaid Services began requiring (1) a shared decision-making (SDM) discussion including use of a patient decision aid and (2) smoking cessation counseling in order to receive reimbursement for LDCT screening. There is little guidance, however, to help healthcare systems implement this requirement. Furthermore, primary care physicians (PCPs) report time constraints, competing demands, and knowledge deficiencies as barriers to optimizing utilization of LDCT screening.

DETAILED DESCRIPTION:
The goal of this study is to create and evaluate an intervention that capitalizes on hospitalization at an urban safety net hospital as an opportunity to connect high risk smokers to lung cancer screening and smoking cessation services. Building on the well-established inpatient tobacco dependence consult service at Boston Medical Center, the investigators will study the effect of adding a nurse-driven LDCT screening SDM intervention to inpatient smoking cessation counseling among screen-eligible hospitalized smokers. Hospitalization may be an ideal time-point for this intervention as it offers 1) a "teachable moment" for patients, when they may be particularly receptive to interventions to reduce smoking-related disease, and 2) an opportunity to offload busy PCPs of the obligation to conduct SDM for LDCT screening.

In Aim 1, screen-eligible patients who are smokers will be randomized into one of the study arms (n=284, 142 per arm) to receive either inpatient 1) SDM (SDM by a thoracic oncology nurse using a decision aid) or 2) usual care and a LDCT informational brochure during inpatient smoking cessation consultation visits. In both arms the thoracic oncology nurse will counsel patients on smoking cessation. The investigators hypothesize that for screen-eligible smokers, inpatient SDM will increase (1) LDCT screening rates, (2) patient knowledge of LDCT screening, and (3) 1 month smoking quit rates compared to usual care.

In Aim 2, the potential for future implementation of the intervention will be evaluated by incorporating stakeholder impressions of the intervention through qualitative interviews. By study end, an inpatient intervention will be created to promote both LDCT screening and smoking cessation among low income and minority smokers. This hybrid study will allow te investigators to establish not only the effectiveness of the intervention, but also help inform future implementation.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized smokers at BMC meeting LDCT screening eligible criteria
* males and females 55-80 years of age
* ≥30-pack years smoking
* current smoker
* able to speak, read, and understand English
* able and willing to participate and provide informed consent

Exclusion Criteria:

* severe co-morbidities expected to limit life expectancy or ability to tolerate surgical resection of a lung cancer, including patients requiring home oxygen therapy (an indicator of severe lung or heart disease), and patients with active cancer
* patients who have already had LDCT screening in the past year

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Completion of LDCT screening | 3 months
  The electronic records review and from the Lung Cancer Screening clinical database created by the Department of Pulmonary Disease and Critical Care at BMC will be reviewed to determine which participants have completed LDCT screening designated as yes or no and if yes the date of the LDCT screening will be recorded..

SECONDARY OUTCOMES:
Knowledge of LDCT screening (experimental group) | Baseline, immediately post SDM, 1 month
  A 21 item instrument developed by Lau and colleagues and modified for a low health literacy population by Crothers will be used. The instrument includes true/false and multiple choice questions that will be used to determine a total score representing knowledge of LDCT screening. The mean percentage of correct responses will be measured so higher scores are better suggesting more knowledge about LDCT screening.
Knowledge of LDCT screening (active comparator group) | Baseline, 1 month
  A 21 item instrument developed by Lau and colleagues and modified for a low health literacy population by Crothers will be used. The instrument includes true/false and multiple choice questions that will be used to determine a total score representing knowledge of LDCT screening.
smoking cessation | 4 weeks
  Dichotomous outcome by self-report of prolonged abstinence at 4 weeks and 7-day point prevalence at 4 weeks, as recommended by the Society for Research on Nicotine and Tobacco and the Russell Standard.

CONTACTS AND LOCATIONS:
Overall Officials: Hasmeena Kathuria, MD, Principal Investigator — Assistant Professor
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kathuria H, Gunawan A, Spring M, Aijaz S, Cobb V, Fitzgerald C, Wakeman C, Howard J, Clancy M, Foreman AG, Truong V, Wong C, Steiling K, Lasser KE, Bulekova K, Wiener RS. Hospitalization as an opportunity to engage underserved individuals in shared decision-making for lung cancer screening: results from two randomized pilot trials. Cancer Causes Control. 2022 Nov;33(11):1373-1380. doi: 10.1007/s10552-022-01620-8. Epub 2022 Aug 23. PMID 35997854